CLINICAL TRIAL: NCT01237522
Title: A Pharmacokinetic Evaluation of Metformin in Relation to the Polymorphism A270S in Healthy Caucasian Volunteers.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Mette Marie Hougaard Christensen, Institute of Public Health, Clinical Pharmacology, University of Southern Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AKF- 377
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2010-06

CONDITIONS: Metformin; Organic Cation Transporter 2; Polymorphism,Single Nucleotide
Keywords: Diabetes Mellitus, Type 2; Metabolic Clearance Rate; Pharmacokinetics; Pharmacogenetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Tolbutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Homozygote for the A270S wildetype (Active Comparator)
  Interventions: Drug: Metformin
- Homo- or heterozygote for A270S minor alleles (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — A single dose study with one tablet of metformin 500 mg, time frame 24 hours
  Other Names: Orabet

SUMMARY:
The aim of the study is to evaluate the pharmacokinetics of metformin in healthy Caucasians volunteers with and without the polymorphism A270S in OCT2,thus the study hypothesis is that renal clearance of metformin is affected in Caucasian with the known single nucleotide polymorphisms A270S in OCT2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Written consent
* rs316019 genotyped
* Age 18-65 years old

Exclusion Criteria:

* Daily medication
* Alcohol abuse
* Pregnancy
* Breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Renal clearance of metformin | 24 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Kim Broesen, Professor, Study Chair — University of Southern Denmark
Locations (1):
- Institute of Public Health, Clinical Pharmacology, University of Southern Denmark, Odense, Denmark